CLINICAL TRIAL: NCT05440318
Title: Exploratory Study to Assess the Use of Wearable Digital Sensors After mRNA Vaccination in Healthy Adults
Brief Title: Use of Wearable Digital Sensors After mRNA Vaccination in Adults
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-CRID-002
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- mRNA Vaccines Recipients: Participants will wear 2 devices during the specified monitoring period. They will wear both a small patch on their chest that captures continuous electrocardiogram (ECG), accelerometry, and temperature data, and a modified smartwatch measuring continuous photoplethysmography (PPG) and accelerometry data.
  Interventions: Device: Wireless wearable digital devices

INTERVENTIONS:
Device: Wireless wearable digital devices — Wireless wearable digital devices (including a small patch, modified watch, and datahub smartphone with electronic Patient Reported Outcomes [ePRO] capability) will be provided to each participant enrolled in the study.

SUMMARY:
The purpose of this study is to explore the physiological and behavioral impact of the immune response to vaccines after receipt of investigational or approved messenger ribonucleic acid (mRNA) vaccines using wearable medical sensors, with the potential of establishing a digital biomarker of vaccine response due to stimulation of the immune system.

DETAILED DESCRIPTION:
Participants will be provided wearable medical sensor equipment and instructions at the start of the study. Participants will have access to device support throughout the study period. The wireless medical devices will be applied prior to vaccination in the concurrent Moderna-sponsored vaccine trial in order to establish an initial baseline of participants' daily physiological patterns.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a concurrent Moderna-sponsored vaccine clinical trial.
* Investigator assessment that participant understands and is willing and physically able to comply with wearing the sensors and follow-up as outlined in the study protocol, including all procedures.
* Participant has provided written informed consent for participation in this study, including all evaluations and procedures as specified in the study protocol.

Exclusion Criteria:

* History of hypersensitivity or allergic reaction to medical adhesive or other history of skin irritation, that, in the opinion of the investigator, contraindicates their use of a wearable medical device.
* Broken skin at the site of wearable location
* Implanted, permanent pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants enrolled in the multi-center, concurrent Moderna-sponsored vaccine trial will be provided the opportunity to enroll in this study. Participants will be screened for eligibility based on their concurrent enrollment in the vaccine trial.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Change From Pre-vaccination Baseline in Heart Rate up to 7 Days After Vaccination | Baseline, up to Day 7
Change From Pre-vaccination Baseline in Respiratory Rate up to 7 Days After Vaccination | Baseline, up to Day 7
Change From Pre-vaccination Baseline in Body Surface Temperature up to 7 Days After Vaccination | Baseline, up to Day 7
Change From Pre-vaccination Baseline in Total Sleep Count Per 24 Hours up to 7 Days After Vaccination | Baseline, up to Day 7
Change From Pre-vaccination Baseline in Moderate to Vigorous Physical Activity Total Minutes Per 24 Hours up to 7 Days After Vaccination | Baseline, up to Day 7
Change From Pre-vaccination Baseline in Digital Biomarker Level up to 7 Days After Vaccination | Baseline, up to Day 7

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Meridian Clinical Research, Lincoln, Nebraska
  - Benchmark Research, Austin, Texas
  - DM Clinical Research- Texas Center for Drug Development, Houston, Texas